CLINICAL TRIAL: NCT01881984
Title: Use of Glycerol Phenylbutyrate (Ravicti™) as a Chaperone to Stabilize Enzyme in Patients With MCAD Deficiency Due to the Common MCAD 985A>G (K304E) Mutation
Brief Title: Use of Ravicti™ in Patients With MCAD Deficiency With the 985A>G (K304E) Mutation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Horizon Pharma Ireland, Ltd., Dublin Ireland (Industry)
Responsible Party: Principal Investigator, Gerard Vockley, MD, PhD, Professor of Pediatrics/Human Genetics, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO13050530
Record Dates: First submitted 2013-06-13; First posted 2013-06-20 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Medium-chain Acyl-CoA Dehydrogenase (MCAD) Deficiency
Keywords: Medium-chain acyl-CoA dehydrogenase deficiency; MCAD deficiency; MCADD; ACADM deficiency; MCADH deficiency; 985A>G mutation; K304E mutation; Ravicti; glycerol phenylbutyrate
MeSH Terms: conditions — Medium chain acyl CoA dehydrogenase deficiency | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ravicti (Experimental): Open Label Study
  Interventions: Drug: Ravicti

INTERVENTIONS:
Drug: Ravicti — Open-label design comparing Ravicti at doses of 2, 4, and 6 grams/m2/day
  Other Names: glycerol phenylbutyrate

SUMMARY:
This is a medical research study to test a medication in adult patients with a disease called medium-chain acyl-CoA dehydrogenase (MCAD) deficiency caused by at least one copy of the 985A>G mutation. The medication is glycerol phenylbutyrate, called Ravicti, which is currently FDA approved for the treatment of urea cycle disorders. Previous research suggests that Ravicti may also be effective in the treatment MCAD deficiency. This study will investigate the safety and efficacy (how well it works) of Ravicti in patients with MCAD deficiency caused by having at least one copy of the 985A>G mutation.

DETAILED DESCRIPTION:
Participation in the study will require one overnight admission and three outpatient visits at the Clinical and Translational Research Center at Children's Hospital of Pittsburgh of UPMC (also called the PCTRC). The total length of the study is 7 weeks.

Subjects will have blood work and an intravenous access line (IV) placed for several blood draws during the visit. Subjects will begin fasting at 8pm during the admission, which means they may consume only non-caloric fluids (water, unsweetened black coffee or tea, or sugar-free beverages). The next morning, fasting blood work will be obtained. The subject can then eat breakfast and will receive the study drug, Ravicti. The total time of fasting will be 12 hours.

Dosing for this study will begin at 2 grams/m2/day, which is about one-fifth (1/5) the dose used for other disorders. The reason for starting the dose lower in MCAD patients is that Ravicti is metabolized by the MCAD enzyme. Following the initial dose, blood will be drawn from the IV every two hours for 8 hours. These blood studies will check the levels of Ravicti in the subject's blood and monitor how the subject's body metabolizes them. The subject will be discharged 8 hours after drug administration. Following discharge, the subject will take Ravicti every day for two weeks.

Visit 2: After two weeks at a dose of 2 grams/m2/day, the subject will fast after 8 PM, and will come to the PCTRC the following morning to have an IV placed and blood draws. If the subject's blood work from the first visit shows that there is no concern, the subject's dose will be increased to 4 grams/m2/day. The subject will receive the first dose at this level in the PCTRC with breakfast, and blood samples will be collected from the IV every 2 hours for the next 8 hours. The subject will continue on this dose for two weeks.

Visit 3: After two weeks at a dose of 4 grams/m2/day, the subject will fast after 8 PM, and will come to the PCTRC the following morning to have an IV placed and blood draws. If the subject's blood work from the previous visit shows that there is no concern, the subject's dose will be increased to 6 grams/m2/day. The subject will receive the first dose at this level in the PCTRC with breakfast, and blood samples will be collected from the IV every 2 hours for the next 8 hours. The subject will continue on this dose for two weeks.

Visit 4 (final): After two weeks at a dose of 6 grams/m2/day, the subject will fast after 8 PM, and will come to the CTRC the following morning to have one blood draw. The subject will return any unused Ravicti, and their study participation will be completed.

All study procedures will be done at no cost to the subjects.

ELIGIBILITY:
Inclusion Criteria:

* confirmation of a diagnosis of MCAD deficiency
* at least one copy of 985A>G MCAD mutation
* ability to follow protocol

Exclusion Criteria:

* positive pregnancy test
* currently breastfeeding
* currently taking any medication for which there is a potential drug interaction with Ravicti, includes corticosteroids, valproic acid, haloperidol, and probenecid
* liver or kidney insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Vockley, MD, PhD, Principal Investigator — University of Pittsburgh/Children's Hospital of Pittsburgh of UPMC
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Kormanik K, Kang H, Cuebas D, Vockley J, Mohsen AW. Evidence for involvement of medium chain acyl-CoA dehydrogenase in the metabolism of phenylbutyrate. Mol Genet Metab. 2012 Dec;107(4):684-9. doi: 10.1016/j.ymgme.2012.10.009. Epub 2012 Oct 18. PMID 23141465
- See also: U.S. National Library of Medicine Genetics Home Reference Information on MCAD Deficiency — http://ghr.nlm.nih.gov/condition/medium-chain-acyl-coa-dehydrogenase-deficiency

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ravicti
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ravicti
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Stress
Description: Changes in the assessments of metabolic stress pre- and post-dosing with Ravicti will be the main outcome variable.
Time Frame: 7 weeks
Population: Due to the small sample size in this Phase I study, details on the analysis cannot be provided due to concerns with subject confidentiality.
Arm/Group | Ravicti
Number analyzed (Participants) | 0

2. Secondary Outcome: Pharmacokinetic (pK)Analysis
Description: Results from the pharmacokinetic (pK)analysis (the rate of conversion of the phenylbutyrate to phenylacetate) will also be reviewed to assess for changes pre- and post-dosing with Ravicti as well as changes in these levels at the different doses of Ravicti.
Time Frame: 7 weeks
Population: as for outcome 1
Arm/Group | Ravicti
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately 7 weeks
Description: The definition of adverse event and a serious adverse event used to collect this information did not differ from the clinicaltrials.gov definition.
Arm/Group | Ravicti
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ravicti (N=4)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Elevated PBA level (Investigations) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Decreased reflexes (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The purpose of this phase 1 trial was to establish a safe dose for treatment of patients with MCAD deficiency due to the common mutations, and to evaluate biomarkers of fatty acid metabolism in treated patients vs their pretreatment values.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes